CLINICAL TRIAL: NCT06527833
Title: Procedure-Specific Approach To Minimize Fistulaization of The Perianal Abscess Cavity After Surgical Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Waleed Ghareeb, Consultant and Lecturer of Surgery, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5697#
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Perianal Fistula
Keywords: perianal abcess; perianal fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non Packing group (Experimental): • In Group (A [Non-Packing group]), The surgery will be performed by making a cruciate incision over the abscess and incision widened using forceps to allow complete drainage of the cavity containing, without any catheter drainage and packing avoided. The lesion will be left open to heal by secondary intension. The patient was advised to have a sitz bath and apply dressing over the cavity.
  Interventions: Procedure: Non Packing of perianal abscess cavity after drainage
- Packing group (Other): In group (B [Packing group]), an elliptical incision will be made, and the abscess will be fully drained then packing the cavity will be done with sterile gauze with a change of dressing every 24 hours until it is completely healed.
  Interventions: Procedure: Packing of perianal abscess cavity after drainage

INTERVENTIONS:
Procedure: Non Packing of perianal abscess cavity after drainage — * All patients will undergo incision and drainage under general anaesthesia.
  * In Group (A [Non-Packing group]), The surgery will be performed by making a cruciate incision over the abscess and incision widened using forceps to allow complete drainage of the cavity containing, without any catheter drainage and packing avoided. The lesion will be left open to heal by secondary intention. The patient was advised to have a sitz bath and apply a dressing over the cavity.
  Arms: Non Packing group
Procedure: Packing of perianal abscess cavity after drainage — an elliptical incision will be made, and the abscess will be fully drained then packing the cavity will be done with sterile gauze with a change of dressing every 24 hours until it is completely healed.
  Arms: Packing group

SUMMARY:
Perianal abscess is a common surgical condition primarily caused by infection of rectal and anal glandular crypts due to non-specific obstruction. Around 10% of cases result from various factors like Crohn's disease, trauma, HIV, STDs, radiation therapy, or foreign bodies. Symptoms include perianal pain, back pain, fever, and more. The main treatment is incision and drainage, but packing during drainage can reduce fistula incidence, though it is associated with pain and cost. Research comparing outcomes with and without packing is limited.

DETAILED DESCRIPTION:
Perianal abscess is a common anorectal condition. Most perianal abscesses are due to infection of the glandular crypts of the rectum and anus caused by non-specific obstruction. A small percentage of cases, around 10%, can be attributed to alternative causes such as Crohn's disease, trauma, human immunodeficiency virus, sexually transmitted diseases, radiation therapy, or foreign bodies.

Perianal abscesses are considered one of the most common colorectal pathologies with an estimated annual incidence of around 20,000 people in Egypt. Perianal abscesses are more common in males as compared to females and more in younger males than older. Also, there is an increased risk of anorectal abscess in conditions such as diabetes, and obesity.

Perianal pain is the most common presentation of perianal abscesses, which may increase with defecation, movement, sitting or coughing. Supra-levator abscesses may present with lower back pain or a dull ache in the pelvic region. Patients may also report fever, malaise, rectal drainage, erythema of surrounding skin and possibly urinary retention. The severity of pain can sometimes prevent the clinician from performing a digital rectal examination or anoscopic examination, therefore if the diagnosis is in doubt, an examination under general anaesthesia should be performed.

Anorectal abscesses can spread into the ischiorectal fossa. They can lead to a horse-shoe-shaped collection or track up towards and through the levator musculature, making management more challenging. Perianal fistulae are a common complication of peri-anal abscesses. Fistulae can be classified according to their tract location in relation to the internal and external sphincters as transphincteric fistula, high intersphincteric fistula, suprasphincteric fistula or extra sphincteric fistula.

In the presence of a perianal fistula, imaging modalities such as CT scans help diagnose intraabdominal pathology such as Crohn's disease and detecting air within the fistulous tract and the abscess cavity. However, MRI is the investigation of choice in evaluating secondary extensions from the fistulous tract and differentiating it from nearby pelvic soft tissue structures.

The management of perianal abscesses is incision and drainage. Without adequately eliminating the source of infection, antibiotics will be ineffective. Minimizing the patient's pain, protecting anal sphincter function and reducing the recurrence of anal fistulae is as important as curing the abscess. Packing at the time of abscess drainage, which requires multiple dressing changes per week for several weeks, can be helpful in providing hemostasis of the inflamed, hypervascular abscess cavity.

However, about 40% of patients with perianal abscess subsequently develop fistula after management. Packing is frequently accompanied by postoperative pain and discomfort, slow wound healing, and increased financial burden yet lower rate of incidence of fistula as demonstrated in Pearce study. Also, there is lack of information comparing postoperative outcomes in managing the perianal abscess cavity with packing and with no packing.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years old with
* perianal abscesses for the first time.

Exclusion Criteria:

* sepsis,
* Previous pelvic radiation
* Pregnancy or lactation
* Immunosuppressive state
* Malignancy
* Refusal to participate will be excluded from this study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Perianal fistula formation | 6 months
  To Compare the incidence of fistulous tract formation in patients drained with non-packing vs. packing approach.
Recurrence of perianal abscess | 6 months
  To Compare the incidence of abscess recurrence formation in patients drained with non-packing vs. packing groups .

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Mostafa Ghareeb, MD, PhD, Principal Investigator — Suez canal University Hospital
Locations (1):
- Suez Canal University Hospital, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No
The IPD will be available and can be provided by the study investigators on reasonable request according to the regulations of our institute.